CLINICAL TRIAL: NCT05380232
Title: Physical Activity and Mortality in Individuals With Type 2 Diabetes: Cross-country Comparison in UK Biobank and China Kadoorie Biobank
Brief Title: Physical Activity and Mortality in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); The Danish Diabetes Association (Other)
Responsible Party: Principal Investigator, Jakob Tarp, Principal Investigator, Aarhus University Hospital
Other Study IDs: 29717
Record Dates: First submitted 2022-05-05; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with type 2 diabetes at the baseline examination: UK Biobank: Prevalent type 2 diabetes is determined by the algorithm of Eastwood et al. (6) or from measured Hba1c ≥48 mmol/mol.
  China Kadoorie Biobank: prevalent type 2 diabetes is based on self-reported current diabetes with a diagnosis age above 30 years, a random plasma blood glucose ≥11.1 mmol/L, or fasting plasma blood glucose ≥7.0 mmol/L.
  Interventions: Behavioral: Leisure-time physical activity

INTERVENTIONS:
Behavioral: Leisure-time physical activity — Self-reported leisure-time physical activity, categorized as; zero (reference), >0-7.49 MET-hrs/week, 7.5-14.9 MET-hrs/week, or ≥15 MET-hrs/week.

SUMMARY:
The primary aim of study is to study the association between leisure-time physical activity and all-cause mortality among individuals with type 2 diabetes in the UK Biobank cohort and the China Kadoorie Biobank cohort. Secondary outcomes are CVD-mortality (both cohorts) and risk of major adverse cardiovascular events (UK Biobank only). Secondary exposures are physical activity from transportation and occupation.

DETAILED DESCRIPTION:
AIM To determine dose-response patterns between leisure-time physical activity and all-cause mortality in individuals with type 2 diabetes in the United Kingdom and China. A secondary aim is to study the association between domain-specific physical activity and all-cause mortality and fatal and non-fatal CVD.

Study design and setting The study is a nested cohort study based on the UK Biobank and China Kadoorie Biobank population-based prospective cohort studies. Both cohorts are designed to study the interrelations between environment, lifestyle, and genes, with the aims of improving the prevention, diagnosis, and treatment of chronic diseases. UK Biobank recruited a total of 502,682 participants (approximately 5.5% of 9.2 million invited) aged 37 to 82 years via 22 assessment centers across England, Wales, and Scotland between 2006 and 2010. At the assessment centers participants completed a touch-screen questionnaire, an interview with a nurse, and a wide variety of physical measurements and biological sampling. A subsample has attended a repeat assessment of all data collected at the baseline examination. Data has been linked with several electronic registries for ongoing follow-up on health status. Ethical approval to establish the UK Biobank cohort was obtained by the North-West Research Ethics Committee and participants gave written informed consent before data collection. China Kadoorie Biobank recruited 515,420 participants aged 30 to 79 years between 2004 and 2008 from 10 regions of mainland China. At the assessment centers participants completed an interviewer-administered questionnaire, physical measurements and provided blood spot tests and non-fasting blood samples. Data has been linked with several electronic registries for ongoing follow-up on health status. China Kadoorie Biobank was approved by the Ethics Committees at Oxford University, the China National Center for Disease Control and from institutional research boards at the local Centers for Disease Control in the 10 included regions.

Study population The Investigators identified individuals with prevalent type 2 diabetes in the UK Biobank from the baseline assessment (2006-2010) and the 1st repeat assessment (2012-2013), and in China Kadoorie Biobank from the baseline assessment (2004-2008).

UK Biobank: Prevalent type 2 diabetes is determined by the algorithm by Eastwood (PMID: 27631769) or from measured Hba1c ≥48 mmol/mol. The algorithm is based on combining information on self-reported diabetes, insulin use, age of diabetes onset, and ethnicity obtained from a questionnaire in addition to self-reported diabetes, self-reported use of medications (see SAP), and age at diabetes diagnosis obtained from an interview with a trained nurse. Both 'probable' and 'possible' type 2 diabetes from the algorithm are included as type 2 diabetes cases. Type I diabetes is removed from the sample by combining information on insulin use, time from diagnosis to initiation of insulin use, and age of diagnosis. These criteria identify 29,236 individuals with type 2 diabetes.

China Kadoorie Biobank: prevalent type 2 diabetes is based on self-reported current diabetes with a diagnosis age above 30 years, a random plasma blood glucose ≥11.1 mmol/L, or fasting plasma blood glucose ≥7.0 mmol/L. These criteria identify 30,300 individuals with type 2 diabetes.

For further detail, please see attached predefined statistical analysis plan (SAP).

ELIGIBILITY:
Inclusion Criteria:

* UK Biobank: Prevalent type 2 diabetes is determined by the algorithm by Eastwood (PMID: 27631769) or from measured Hba1c ≥48 mmol/mol.
* China Kadoorie Biobank: Self-reported current diabetes with a diagnosis age above 30 years, a random plasma blood glucose ≥11.1 mmol/L, or fasting plasma blood glucose ≥7.0 mmol/L

Exclusion Criteria:

* None

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: See statistical analysis plan
Sampling Method: Non-Probability Sample
Enrollment: 502682 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Through longest available follow-up, up to 14.5 years (UK Biobank)
  Mortality status optained from registries. The longest available follow-up from baseline examination will be used. Deaths during the first 3 years will be left-censored.
All-cause mortality | Through longest available follow-up, up to 12.4 years (China Kadoorie Biobank)
  Mortality status optained from registries. The longest available follow-up from baseline examination will be used. Deaths during the first 3 years will be left-censored.

SECONDARY OUTCOMES:
Cardiovascular mortality | Through longest available follow-up, up to 14.5 (UK Biobank) and 0.4 (China Kadoorie Biobank) years
  Cardiovascular mortality status optained from registries (I00 to I-99). The longest available follow-up from baseline examination will be used. Deaths during the first 3 years will be left-censored.
Major adverse cardiovascular events (MACE) | Through longest available follow-up, up to 14.5 (UK Biobank only)
  MACE status optained from registries (I20-I25, I60, I61, I63, or I64 in addition to cardiovascular mortality). The longest available follow-up from baseline examination will be used. Participants with events during the first 3 years will be left-censored.

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT05380232/SAP_000.pdf